CLINICAL TRIAL: NCT03952273
Title: Randomized Clinical Comparison of the Combined Sirolimus Eluting and Endothelial Progenitor Cell Combo™ Stent and the Biolimus Eluting Absorbable Polymer Coated BioMatrix Alpha™ Stent in Patients Treated With Percutaneous Coronary Intervention.
Brief Title: Sort Out XI - Combo Stent Versus BioMatrix Alpha Stent
Acronym: SORTOUTXI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phillip Freeman (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); OrbusNeich (Industry); Biosensors International (Other)
Responsible Party: Sponsor-Investigator, Phillip Freeman, Principal Investigator, MD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sort Out XI
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: Drug eluting stent; Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combo (Active Comparator): PCI with COMBO stent
  Interventions: Combination Product: PCI with Combo™ stent
- BioMatrix Alpha (Active Comparator): PCI with BioMatrix Alpha stent
  Interventions: Combination Product: PCI with BioMatrix Alpha™ stent

INTERVENTIONS:
Combination Product: PCI with BioMatrix Alpha™ stent — Randomozation between either Sirolimus eluting and endothelial progenitor cell Combo™ stent or Biolimus eluting absorbable polymer coated BioMatrix Alpha™ stent
  Other Names: Biolimus eluting absorbable polymer coated BioMatrix Alpha™ stent
  Arms: BioMatrix Alpha
Combination Product: PCI with Combo™ stent — Randomozation between either Sirolimus eluting and endothelial progenitor cell Combo™ stent or Biolimus eluting absorbable polymer coated BioMatrix Alpha™ stent
  Other Names: Combined sirolimus eluting and endothelial progenitor cell Combo™ stent
  Arms: Combo

SUMMARY:
SORT OUT XI Comparison of Combo™ stent and BioMatrix Alpha™ stent in the treatment of unselected patients with ischemic heart disease.

DETAILED DESCRIPTION:
Randomized clinical comparison of the Sirolimus eluting and endothelial progenitor cell Combo™ stent and the Biolimus eluting absorbable polymer coated BioMatrix Alpha™ stent in patients treated with percutaneous coronary intervention

ELIGIBILITY:
Inclusion Criteria:

All patients aged ≥18 years who are eligible for treatment with one or several drug-eluting coronary stents at one of the three heart centers in Aarhus, Odense and Aalborg can be included in the study.

Exclusion Criteria:

* Age < 18 years
* The patient does not wish to participate
* The patient is not able to consent to randomization (eg. intubated patients)
* The patient do not speak Danish
* The patient is already included in the SORT OUT XI study
* Life expectancy <1 year
* Allergic to study related treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3141 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Device-related Target Lesion Failure (TLF) The composite of cardiac death, target-vessel myocardial infarction (MI), or ischemia-driven target-lesion revascularization | Within 12 months
  The primary endpoint will be analyzed using the Kaplan-Meier method. Hazard ratios between groups will be calculated using a Cox proportional hazard model and the primary endpoint in the two per protocol treated groups will be compared with an upper one-sided 95% confidence interval. Patients treated with the ComboTM stent will be used as the reference group.
Target Lesion Revascularisation (TLR) | Within 12 months
  Repeat/new revascularization (PCI or CABG) within the stent or within a 5-mm border proximal or distal to the stent. (Angina, CCS > 1 related to the index lesion/vessel and diameter stenosis ≥ 50%. Diameter stenosis will be assessed by eyeballing, FFR <0.80, or iFR< 0.90). TLR will be clinically driven.

SECONDARY OUTCOMES:
Individual components of the primary end point comprise the secondary end points | Clinical follow-up will be continued through 5 years
  cardiac death; MI; clinically indicated TLR; all death (cardiac and noncardiac) and target vessel revascularisation (TVR); definite, probable, possible, and overall stent thrombosis according to the Academic Research Consortium definition (22); and a patient-related composite end point (all death, all MI (including procedure related MI), or any revascularization). For continuous variables, the difference between the treatment groups will be evaluated using Wilcoxon's rank-sum test. For discrete variables, the differences will be given as numbers and in percentages and will be analyzed using Fisher's exact test. Two-sided test will be used, and a pvalue of 0.05 considered significant.
Number of participants with Cardiac Death | Through 5 years
Number of participants with Myocardial Infarction | Through 5 years
  The acute MI diagnosis follows "The Joint ESC/ACCF/AHA/WHF Task Force on "Third Universal Definition of MI" (23), which has been adapted by Academy Research Consortium (22).
  In cases of updates of the definition of MI, the latest definition will be used.
Target Lesion Revascularization due to clincal symptoms | Through 5 years
  Angina, CCS > 1 related to the index lesion/vessel and diameter stenosis ≥ 50%. Diameter stenosis will be assessed by eyeballing, FFR <0.80, or iFR< 0.90.
Number of patients with all cause mortality | Through 5 years
  Cardiac and non-cardiac
Target Vessel Revascularization due to clincal symptoms | Through 5 years
  Angina, CCS > 1 related to the index lesion/vessel and diameter stenosis ≥ 50%. Diameter stenosis will be assessed by eyeballing, FFR <0.80, or iFR< 0.90.
Number of patients with stent thrombosis | Through 5 years
  Definite, probable, possible and overall according to the Academic Research Consortium definition (22)
Number of patients with Patient-related composite end point | Through 5 years
  All death, all MI (including procedure related MI) or any revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Freemann, MD, Principal Investigator — Aalborg University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Skejby, Aarhus
  - Odense Unversity Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
Only shared with collaborators

REFERENCES:
- [Derived] Eftekhari A, Jensen LO, Veien K, Raungaard B, Rasmussen JG, Maeng M, Terkelsen CJ, Ellert-Gregersen J, Stottrup NB, Lassen JF, Hansen HS, Thim T, Jensen RV, Nielsen R, Jensen SE, Kristensen SD, Hougaard M, Junker A, Christensen MK, Aaroe J, Froslev T, Jakobsen L, Christiansen EH. Biolimus-Eluting Biomatrix Stent vs a Dual-Therapy Sirolimus-Eluting Stent in PCI: The SORT OUT XI Randomized Trial. J Am Coll Cardiol. 2025 Jul 15;86(2):106-115. doi: 10.1016/j.jacc.2025.05.012. Epub 2025 May 21. PMID 40406942
- [Derived] Eftekhari A, Christiansen EH, Lassen JF, Raungaard B, Jakobsen L, Jensen LO. Randomized comparison of the combined Sirolimus eluting and endothelial progenitor cell combo Stent vs. biolimus eluting absorbable polymer coated biomatrix alpha stent in patients undergoing percutaneous coronary intervention: Rationale and study design of the Scandinavian Organization for randomized trials with clinical outcome (SORT OUT) XI trial. Am Heart J. 2025 May;283:37-42. doi: 10.1016/j.ahj.2025.01.012. Epub 2025 Jan 25. PMID 39870125